CLINICAL TRIAL: NCT01074268
Title: NN1250-3585: A Trial Investigating the Efficacy and Safety of NN1250 Compared to Insulin Detemir in Subjects With Type 1 Diabetes Mellitus in a Basal/Bolus Treatment Regimen / NN1250-3725: An Extension Trial to NN1250-3585 Investigating Safety and Efficacy of NN1250 Compared to Insulin Detemir in Subjects With Type 1 Diabetes Mellitus in a Basal/Bolus Treatment Regimen (BEGIN™: BB T1)
Brief Title: Comparison of NN1250 Plus Insulin Aspart With Insulin Detemir Plus Insulin Aspart in Type 1 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3585; 2009-011672-29 (EudraCT Number); U1111-1111-7249 (Other: WHO); JapicCTI-101067 (Registry Identifier: JAPIC); 2009-015721-36 (EudraCT Number); U1111-1114-9479 (Other: WHO); JapicCTI-22-0677 (Registry Identifier: JAPIC); NCT01190956 (obsolete NCT alias)
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IDet (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Injected s.c. (under the skin) once daily. Dose was individually adjusted.
  Arms: IDeg OD
Drug: insulin detemir — Injected s.c. (under the skin) once daily or twice daily (BID). Dose was individually adjusted.
  Arms: IDet
Drug: insulin aspart — Injected s.c. (under the skin) as mealtime insulin. Dose was individually adjusted.

SUMMARY:
This trial is conducted in Asia, Europe, Japan and South America. The aim of the trial is to compare the efficacy, safety and tolerability of NN1250 (insulin degludec ([Deg]) with insulin detemir (IDet), both combined with insulin aspart.

The main period is registered internally at Novo Nordisk as NN1250-3585 while the extension period is registered as NN1250-3725.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 12 months
* Current treatment with any basal bolus insulin for at least 12 months
* HbA1c below or equal to 10.0%
* Body Mass Index (BMI) below or equal to 35.0 kg/m^2
* For Japan only: Minimum age is 20 years
* For the extension trial only: Completed the six-month treatment period in trial NN1250-3585 (NCT01074268)

Exclusion Criteria:

* Use of any other antidiabetic drug than insulin within the last 3 months
* Cardiovascular disease within the last 6 months
* Uncontrolled treated/untreated severe hypertension
* Recurrent severe hypoglycemia or hypoglycemic unawareness or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures
* Cancer and medical history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (64):
- Argentina (4):
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Ciudad Autónoma de Bs As
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Rosario
- Brazil (5):
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Marília
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, São Paulo
- Finland (7):
  - Novo Nordisk Investigational Site, Hämeenlinna
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Seinäjoki
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- India (9):
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Ahmedabad
  - Novo Nordisk Investigational Site, Bilāspur
  - Novo Nordisk Investigational Site, Dhantoli, Nagpur
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, New Dehli
  - Novo Nordisk Investigational Site, Ramdaspeth / Nagpur
  - Novo Nordisk Investigational Site, Thriruvananthapuram
- Italy (11):
  - Novo Nordisk Investigational Site, Bari
  - Novo Nordisk Investigational Site, Forlì
  - Novo Nordisk Investigational Site, Gazi
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Olbia
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Partinico
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Torino
  - Novo Nordisk Investigational Site, Treviglio
  - Novo Nordisk Investigational Site, Treviso
- Japan (13):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi
  - Novo Nordisk Investigational Site, Imizu-shi
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Yokohama
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- United Kingdom (14):
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Carmarthen
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Penarth
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Torquay
  - Novo Nordisk Investigational Site, Wirral, Merseyside

REFERENCES:
- [Result] Davies MJ, Gross JL, Ono Y, Sasaki T, Bantwal G, Gall MA, Niemeyer M, Seino H; BEGIN BB T1 Study Group. Efficacy and safety of insulin degludec given as part of basal-bolus treatment with mealtime insulin aspart in type 1 diabetes: a 26-week randomized, open-label, treat-to-target non-inferiority trial. Diabetes Obes Metab. 2014 Oct;16(10):922-30. doi: 10.1111/dom.12298. Epub 2014 May 8. PMID 24702700
- [Result] Davies M, Sasaki T, Gross JL, Bantwal G, Ono Y, Nishida T, Tojjar D, Seino H. Comparison of insulin degludec with insulin detemir in type 1 diabetes: a 1-year treat-to-target trial. Diabetes Obes Metab. 2016 Jan;18(1):96-9. doi: 10.1111/dom.12573. Epub 2015 Oct 19. PMID 26435472
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 55 sites in 7 countries: Brazil (2), Finland (8), India (10), Italy (6), Japan (15), Macedonia (1) and United Kingdom (13). For the extension trial, one trial site in Italy did not enroll any subject since approval was not obtained before the start of the trial from the IEC.
Pre-assignment Details: All subjects who completed the 26-week main trial (NN1250-3585, NCT01074268) and were found to be eligible for the extension trial were offered to participate in the 26-week extension trial (NN1250-3725). The total duration of treatment was 52 weeks (26 weeks + 26 weeks), separated by 1 week of follow-up from the main trial.
Groups:
- IDeg OD: Insulin degludec (IDeg) was given subcutaneously (s.c.) once daily (OD) in the evening in combination with insulin aspart (IAsp) as meal-time insulin. IDeg OD was given for 26 weeks in the main period and for another 26 weeks in the extension period.
- IDet OD: Insulin detemir (IDet) was given subcutaneously (s.c.) once daily (OD) in the evening or twice daily (BID) morning and evening in combination with insulin aspart (IAsp) as meal-time insulin. IDet was given for 26 weeks in the main period and for another 26 weeks in the extension period.
Period: Main: Week 0 to 26 (NN1250-3585)
Arm/Group | IDeg OD | IDet OD
Started | 303 | 153
Full Analysis Set | 302 (One subject was withdrawn because the subject was randomised in error (screening failure)) | 153
Exposed | 301 (Two subjects withdrew prior to exposure to trial drugs) | 152 (One subject withdrew prior to exposure to trial drugs)
Completed | 283 | 138
Not Completed | 20 | 15
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal criteria | 6 | 3
Not completed — Unclassified | 8 | 5
Period: Extension: Week 27 to 52 (NN1250-3725)
Arm/Group | IDeg OD | IDet OD
Started | 248 (Thirty five subjects from main trial did not continue into the extension) | 122 (Sixteen subjects from main trial did not continue into the extension)
Completed | 242 | 115
Not Completed | 6 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal criteria | 2 | 2
Not completed — Unclassified | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD | IDet OD | Total
Number analyzed (Participants) | 302 | 153 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (14.9) | 41.7 (14.4) | 41.3 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 67 | 219
  Male | 150 | 86 | 236
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.0 (1.0) | 8.0 (0.9) | 8.0 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.9 (4.0) | 9.5 (4.0) | 9.8 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Main Trial (Primary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 26 Weeks of Treatment
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 302 | 153
percentage of glycosylated haemoglobin | -0.73 (0.88) | -0.65 (0.86)

2. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment
Time Frame: Week 0, Week 52
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 302 | 153
percentage of glycosylated haemoglobin | -0.46 (0.93) | -0.47 (0.88)

3. Secondary Outcome: Main Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 26
Description: Mean of 9-point self-measured plasma glucose profile (SMPG) after week 26. Plasma glucose was measured before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before main evening meal, 90 minutes after the start of main evening meal, before bedtime, at 04:00 AM and before breakfast on the following day.
Time Frame: Week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 5 subjects, all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 299 | 151
mmol/L | 7.9 (2.1) | 7.8 (1.9)

4. Secondary Outcome: Extension Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 52
Description: Mean of 9-point self-measured plasma glucose profile (SMPG) at week 52. Plasma glucose was measured before breakfast, 90 minutes after the start of breakfast, before lunch, 90 minutes after the start of lunch, before main evening meal, 90 minutes after the start of main evening meal, before bedtime, at 04:00 AM and before breakfast on the following day.
Time Frame: Week 52
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF. For 4 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 150
mmol/L | 7.8 (1.9) | 7.8 (2.0)

5. Secondary Outcome: Main Trial (Secondary Endpoint): Change in Fasting Plasma Glucose (FPG) After 26 Weeks of Treatment
Description: Change from baseline in FPG after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 6 subjects change in FPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 148
mmol/L | -2.60 (4.87) | -0.62 (4.49)

6. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Fasting Plasma Glucose (FPG) After 52 Weeks of Treatment
Description: Change from baseline in FPG after 52 weeks of treatment
Time Frame: Week 0, Week 52
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF. For 6 subjects change in FPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 148
mmol/L | -2.19 (4.99) | -0.82 (4.79)

7. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes: episodes requiring active assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes: episodes where the subject was able to treat her/himself and plasma glucose below 3.1 mmol/L, with or without symptoms.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 152
Episodes/100 years of patient exposure | 4583 | 4569

8. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes: episodes requiring active assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes: episodes where subject was able to treat her/himself and plasma glucose below 3.1 mmol/L, with or without symptoms. Nocturnal hypoglycaemic episodes are defined as occuring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 152
Episodes/100 years of patient exposure | 414 | 593

9. Secondary Outcome: Extension Trial (Secondary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes: episodes requiring active assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes: episodes where the subject was able to treat her/himself and plasma glucose below 3.1 mmol/L with or without symptoms
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator in the main trial including subjects carried through to the extension trial.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 152
Episodes/100 years of patient exposure | 3778 | 3926

10. Secondary Outcome: Extension Trial (Secondary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: as for outcome 8
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: as for outcome 9
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 152
Episodes/100 years of patient exposure | 338 | 481

11. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Treatment Emergent Adverse Events (AEs)
Description: Rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no/transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect or important medical issues
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: as for outcome 9
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDeg OD | IDet OD
Number analyzed (Participants) | 301 | 152
Events/100 years of patient exposure
  Adverse events (AEs) | 459 | 420
  Serious AE | 20 | 17
  Severe AE | 23 | 35
  Moderate AE | 48 | 45
  Mild AE | 388 | 341
  Fatal AE | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 52 weeks + 7 days follow up
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg OD | IDet OD
Serious Adverse Events (participants affected / at risk) | 36/301 | 11/152
Other Adverse Events (participants affected / at risk) | 185/301 | 89/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=301) | IDet OD (N=152)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exocrine pancreatic function test abn (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (16) | 5 (8)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 9 (9) | 5 (6)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 4 (4) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=301) | IDet OD (N=152)
Nasopharyngitis (Infections and infestations) | 94 (162) | 49 (79)
Upper respiratory tract infection (Infections and infestations) | 34 (61) | 17 (28)
Hypoglycaemia (Metabolism and nutrition disorders) | 15 (25) | 11 (13)
Headache (Nervous system disorders) | 42 (84) | 12 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 8 (12)
Diabetic retinopathy (Eye disorders) | 20 (22) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 20 (25) | 9 (10)
Pyrexia (General disorders) | 16 (24) | 9 (10)
Gastroenteritis (Infections and infestations) | 22 (23) | 10 (11)
Influenza (Infections and infestations) | 14 (14) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (24) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.